CLINICAL TRIAL: NCT02513238
Title: Mesenchymal Stem Cells for Radiation-induced Xerostomia (MESRIX) in Previous HPV-positive Oropharyngeal Head and Neck Cancer Patients - A Safety and Feasibility Study
Brief Title: Mesenchymal Stemcells for Radiation Induced Xerostomia
Acronym: MESRIX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Christian Grønhøj Larsen, MD, PhD student, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1406653
Record Dates: First submitted 2015-07-02; First posted 2015-07-31 (Estimated); Results first posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-11

CONDITIONS: Xerostomia
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stemcells injected into submandibularis (Active Comparator): The surgical procedure is done under local anaesthesia using ultrasonic guidance and sterile technique. After receiving the MSC-suspension , the surgeon will identify the submandibular glands and inject the suspension MSCs into the submandibular gland. Calculation of injected number of MSCs pr. participant rests on the following calculation: 2.8 x 10^6 MSC / Cm^3 X volume , where volume is the volume of the submandibular gland, and a gland-volume of app. 7-8cm3 is the norm. Therefore the amount of cells given to each participant will be app. 4.6 x 10^7 MSC in total. Afterwards the participant will be given a band-aid and over the counter analgesics.
  Interventions: Drug: Mesenchymal stem cell
- Saltwater injected into submandibularis (Placebo Comparator): The surgical procedure is done under local anaesthesia using ultrasonic guidance and sterile technique. After receiving the placebo-suspension , the surgeon will identify the submandibular glands and inject the suspension. Placebo will be 2ml of Isotonic NaCl (0,9mg/ml) and HA 1%.
  Interventions: Drug: Isotonic NaCl

INTERVENTIONS:
Drug: Mesenchymal stem cell — Stemcells injected into submandibularis
  Arms: Stemcells injected into submandibularis
Drug: Isotonic NaCl
  Arms: Saltwater injected into submandibularis

SUMMARY:
The current study aims to assess the safety and feasibility of the injection of autologous adipost tissue derived MSCs on radiation-induced salivary gland hypofunction and xerostomia in head and neck cancer participants. The project can potentially help to develop a clinically relevant treatment option for the growing number of patients suffering from xerostomia after radiotherapy. The development of new therapies is especially important, since only sub-optimal symptomatic treatments are currently available and the symptom of xerostomia greatly reduces the quality of life.

DETAILED DESCRIPTION:
Design Randomized, controlled trial with blinding. To maintain allocation concealment all participants, care givers, trial investigators and outcome assessors except the Blood Bank staff will be blinded to the intervention. Staff from the Blood Bank will not have direct contact with the patients (hereafter the participants) as such.

Project plan For inclusion in the study participants will have their usual medical history taken according to guidelines from the Ear, Nose and Throat Surgical Department, Copenhagen University Hospital Rigshospitalet.

All participants will undergo a mini lip-suction, from which MSCs will be ex vivo expanded in a good manufacturing practice (GMP)-approved clean room facility (The Blood Bank, section 2014). When the cells arrive at the Blood Bank, participants will be randomized to either ex vivo expansion of their mesenchymal stem cells or having them frozen for potential later use. Expected ex vivo expansion phase is 3-4 weeks. The purification and isolation will be based on a protocol previously approved for clinical use.

Amount of MSCs required for injection Based on published animal studies the amount given for xerostomia to mice varies from 2 x 105 to 2 x 106 [19]. To convert these mice data to a realistic dose in humans we have extrapolated based on the following data: The volume density of submandibular glands very closely approximates 1 (1.06-1.07 mg/mm3) [27]. In the mice studies on radiotherapy the mean gland weight was approximately 350mg, which corresponds to an approximate volume of 350mm3. Therefore the mouse dose pr. gland volume is approximately 286.000-2.860.000cells pr. cm3 gland (when calculated from either 1 x 105 to 1 x 106). The volume of the submandibular gland in human subjects after radiotherapy is 6.6-7.9cm3 [28]. This corresponds to an approximate dose pr. patient of between 1.9 x 106 to 2.2 x 106, or 1.9 x 107 to 2.2 x 107 cells pr. submandibular gland. From the above assumptions and in order not to give to few cells we have chosen to proceed with the maximum dose corresponding to 2.8*10^6 MSC/cm^3 gland, i.e. a maximum total dose per patient of approximately 4,6 * 10^7 MSCs. However to standardize the dose given to patients, the amount given will be standardized to the size of their submandibular glands, as described below.

Injection of MSCs into submandibular glands Subjects will go to the ENT-department, section 2073 for inpatient procedures. The surgical procedure is done under local anaesthesia using ultrasonic guidance and sterile technique. After receiving the MSC-suspension or placebo-suspension, the surgeon will identify the submandibular glands and inject the suspension MSCs. Calculation of injected number of MSCs pr. participant rests on the following calculation: , where volume is the volume of the submandibular gland, and a gland-volume of app. 7-8cm3 is the norm. Therefore the amount of cells given to each participant will be app. in total. Afterwards the participant will be given a band-aid and over the counter analgesics. The MSCs will be suspended in Isotonic NaCl (0,9 mg/ml) and Human Albumin (HA) 1% to a final volume of 2ml. Placebo will be 2ml of Isotonic NaCl (0,9mg/ml) and HA 1%.

Follow-up MRI of the recipient place will be performed after 3-4 weeks and 3-4 months postoperatively. MRI is used for volume determination of salivary glands and control of recipient place.

After 3-4 months, a small biopsy is randomly taken from one of the two salivary glands. The procedure takes place under local anaesthesia. Histology is determined (samples are blinded to the pathologist).

When the final MRI, biopsy and salivary function test has been performed approx. 3-4 months after treatment specific study related tests and activities are concluded. To detect late complications or late adverse events all study participants who received MSC-treatment are invited for a check-up 1 year and 3 years after treatment.

Safety, isolation and propagation of MSC The Blood Bank has its cell-tissue approval from the Danish Health and Medicines Authority (according to the Danish Tissue Law), as well as a Manufacturer's/Importer's Authorisation regarding Human Medicinal Products, the necessary physical facilities, personnel and operational resources to produce MSCs in accordance with good manufacturing practice (GMP).

The MSC product will be tested for recognized surface markers (CD73, CD90, CD105,) using flow cytometry, and undergo general quality checks before the final release (cell viability and tests for microorganisms). With regard to the cultivation of the MSC we will use basal medium supplemented with human platelet lysate from healthy blood donors instead of the former use of animal-derived serum (fetal bovine serum, FBS). This has the following benefits: 1) No likelihood of transfection of both known and unknown animal pathogens, or risk of xeno-immunization 2) Small batch-to-batch variation and thus more consistent growth performance, since each group is prepared from approx. 50 healthy donors.

All harvest, isolation, expansion, etc. of MSC will be in accordance with GMP regulations. The Blood Bank has clean room facilities approved by the Danish Health and Medicines Authority for GMP compliant cell expansion for clinical use, and all studies will be carried out by specially trained personnel.

Assessment of xerostomia and subjective treatment outcome The subjective effect of the treatment is assessed by a 100 mm visual analogue scale of xerostomia filled out by the patient [31] and a physician-rated questionnaire [32], both carried out before as well as after treatment. Each participant will also be asked about daily symptoms of dry mouth according to the UKU side-effect rating scale item 3.3 [29]. This scale includes four scores where 0 denotes no feeling of dry mouth, 1 denotes a slight feeling of dry mouth, 2 denotes a severe feeling of dry mouth, and 3 denotes troublesome feeling of dry mouth that makes speech and eating difficult.

Assessment of salivary flow rate and objective treatment outcome Changes in the secretion rate of the unstimulated whole saliva in the oral cavity is probably the most important parameter for the biological development of xerostomia and accompanying pathological oral conditions. Whole saliva, e.g., the mixed secretions from the major and minor salivary glands is mixed in the oral cavity. A correct determination of this value is crucial for the assessment of treatment outcome in this project. For assessment of the saliva flow rate, whole saliva will be collected between 9 and 12 a.m. Subjects will refrained from eating, drinking, smoking and oral hygiene for 2 hr before the collection. After being seated upright in a chair, they relax for 5 min and are then instructed to make as few movements as possible, including swallowing, during the collection.

Before and after treatment unstimulated whole saliva will be collected using the spitting method [33] where participants spit their saliva into a collection container over a period of 15 minutes. The salivary flow rate (SFR) (ml / min) is determined as the increase in weight of the container divided by the collection time in minutes.

After the collection of unstimulated saliva, the subjects are instructed to chew on 1 g of sterile paraffin wax. They will be asked to keep their mouths closed during chewing and to avoid swallowing. Every 60 sec they will be asked to spit into a new saliva collector before starting a new chewing period. This will be repeated for 5 min.

To assess treatment outcome of the submandibular glands, saliva is also collected directly from the floor of the mouth in an unstimulated and stimulated state. The unstimulated whole saliva flow rate of the submandibular glands will be assessed by the swab method with cotton rolls placed buccally in each maxillary molar region and under the tongue on the floor of the mouth. Immediately prior to the start of collection they will be asked to swallow, in case this is not possible saliva will be extracted by a pipette. Collection takes place during two subsequent periods of 3 min and, at the end of each period, the chin and lips will be wiped with a napkin. Saliva flow rates are determined by weight (1 g equals 1 ml of saliva) with rolls and napkins weighed before collection and reweighed after. The flow rates is calculated as the increment in weight during collection and expressed as millilitres per minute. Saliva from the cotton rolls will be extracted by centrifugation (1500g) and analyzed for its composition. This stimulated collection process will be performed afterwards with citrus-containing rolls to stimulate the submandibular glands maximally. From each of these collections of saliva, saliva will be aliquoted and stored at -800C.

Chemical analysis of saliva Whole saliva contains a large number of bacteria and epithelial cells, as well as gingival crevicular fluid. Therefore, whole saliva is normally not suited for the analysis of sensitive chemical parameters. For this purpose, the selectively collected saliva from individual glands is much better. As a result, the majority of analyzes can be performed from either the parotid and submandibular gland / sublingualis saliva. The following analyzes will be performed on the collected saliva: pH and bicarbonate by ionic balance estimation [34], sodium, potassium, calcium, phosphate, chloride and fluoride [35], total protein and selected proteins [36] and amylase [37]. The purpose of the studies is to evaluate whether saliva will be normalized after treatment, and thus provide an estimate of the saliva dental and mucosal protective capacity before and after treatment.

Data collection and analysis Source data: There will be source documentation for all data in Case Report Form (CRF).

The study director allows direct access to study data and study documents for the monitoring, audit and inspection of the Science Ethics Committee, the Danish Health and Medicines Authority or similar authorities in other countries. Permission will be sought from the DPA for the processing of personal data under the Danish Data Protection Act. Applications will be sent via the legal secretariat, Rigshospitalet.

ELIGIBILITY:
Inclusion Criteria:

Previous radiotherapy for HPV-positive oropharyngeal head and neck cancer with bilateral irradiation of the neck.

* 2 years follow-up without recurrence
* Clinically reduced salivation and hyposalivation, evaluated by a screening
* Unstimulated salivary flow rate between less than 0.2ml/min and above 0.05ml/min
* Only participants with previous T1-T2 and N0, N1 or N2a.
* Informed consent
* Grade 1-3 xerostomia as evaluated by the UKU side effect rating scale

Exclusion Criteria:

* Any cancer in the previous 2 years
* Xerogenic medications
* Any other diseases of the salivary glands, e.g. Sjögrens syndrome, sialolithiasis, etc.
* Pregnancy or planned pregnancy within the next 2 years
* Breastfeeding
* Any other disease/condition judged by the investigator to be grounds for exclusion
* Treatment with anticoagulant that cannot be stopped during the intervention period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08-08 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

REFERENCES:
- [Derived] Gronhoj C, Jensen DH, Glovinski PV, Jensen SB, Bardow A, Oliveri RS, Specht L, Thomsen C, Darkner S, Kiss K, Fischer-Nielsen A, von Buchwald C. First-in-man mesenchymal stem cells for radiation-induced xerostomia (MESRIX): study protocol for a randomized controlled trial. Trials. 2017 Mar 7;18(1):108. doi: 10.1186/s13063-017-1856-0. PMID 28270226

RESULTS

PARTICIPANT FLOW:
Groups:
- Saltwater Injected Into Submandibularis: The surgical procedure is done under local anaesthesia using ultrasonic guidance and sterile technique. After receiving the placebo-suspension , the surgeon will identify the submandibular glands and inject the suspension. Placebo will be 2ml of Isotonic NaCl (0,9mg/ml) and HA 1%.
  Isotonic NaCl
Period: Overall Study
Arm/Group | Stemcells Injected Into Submandibularis | Saltwater Injected Into Submandibularis
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stemcells Injected Into Submandibularis | Saltwater Injected Into Submandibularis | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 60 [45 to 65] | 60 [40 to 65] | 60 [40 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 10 | 10 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety
Description: Criteria for Adverse Events (CTCAE). Since this is a local treatment with MSCs the primary safety measures are: All measures of adverse events will be graded according to Common Terminology
Time Frame: 4 months
Measure: Number; unit: participants
Arm/Group | Stemcells Injected Into Submandibularis | Saltwater Injected Into Submandibularis
Number analyzed (Participants) | 15 | 15
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Stemcells Injected Into Submandibularis | Saltwater Injected Into Submandibularis
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT02513238/Prot_SAP_000.pdf